CLINICAL TRIAL: NCT03646591
Title: Pilot Study on Feasibility and Safety of FLOT Regimen as Neoadjuvant Chemotherapy in Chinese Gastric Cancer Patients
Brief Title: Feasibility and Safety of Neoadjuvant Chemotherapy (FLOT ) for Gastric Cancer Patients in China
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BIRENDRA KUMAR SAH, Surgeon, Ruijin Hospital
Other Study IDs: Dragon III- Pilot study
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Chemotherapy Effect
Keywords: gastric cancer; neoadjuvant chemotherapy; FLOT regimen
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant chemotherapy: FLOT Chemotherapy regimen
  A cycle consist of Day 1: 5-fluorouracil (5-FU) 2600mg/M2 intravenous Via peripherally inserted central catheter (PICC) for 24 hour Day 1: Leucovorin 200mg/M2 intravenous Day 1: Oxaliplatin 85mg/ M2 intravenous Day 1: Docetaxel 50mg/M2 intravenous Repeated every 15th day
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Patients will receive four cycles of the standard dose of FLOT chemotherapy prior to curative gastrectomy. And four cycles of the FLOT chemotherapy is recommended after surgery. Preventive antiemetic and dexamethasone are allowed before chemotherapy, growth factor, or other supportive medicines are allowed for treatment only. Surgical intervention is allowed for acute bleeding or other surgical emergencies.
  Other Names: FLOT

SUMMARY:
Neoadjuvant chemotherapy for advanced-stage gastric cancer is justified by various studies, however, there was not any large scale randomized controlled trial (RCT) to support it until German oncologist introduced a novel regimen(FLOT regimen) in 2017. Investigator assessed the FLOT regimen for safety and feasibility in Chinese gastric cancer patients.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy for advanced-stage gastric cancer is justified by various studies, however, there was not any large scale RCT to support it until German oncologist introduced a novel regimen(FLOT regimen) in 2017. FLOT regimen was prescribed for German patients and various questions are raised by experts from Eastern countries. As the FLOT regimen was officially included in NCCN 2018 guidelines, the investigator used standard protocol of FLOT regimen on Chinese gastric cancer patients. Safety and feasibility were assessed carefully to provide basic data for further large scale studies in China.

ELIGIBILITY:
Inclusion Criteria:

* Sex: all
* Histology confirmed adenocarcinoma of the stomach or esophagogastric junction.
* Clinical stage: Clinical Tumor-Node-Metastasis (cTNM): stage III，IVa
* Performance status: Eastern Cooperative Oncology Group ECOG 0- 2
* Adequate renal, hepatic, hematologic, and pulmonary function.
* Written informed consent

Exclusion Criteria:

* Uncontrolled cardiac disease, or other clinically significant uncontrolled comorbidities
* Distant metastases
* Prior chemo or radiotherapy
* Inclusion in another clinical trial
* Known contraindications or hypersensitivity for planned chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of operable gastric cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Completion rate of preoperative FLOT regimen | upto 3 months
  How many patients completed the plan preoperative chemotherapy regimen

SECONDARY OUTCOMES:
Adverse events | Upto three months
  Chemotherapy related adverse events according to the CTCAE version 3.0
Pathological response rate | Upto three months
  According to tumor regression grading(TRG)
Postoperative morbidity | Upto one month after hospital discharge
  Postoperative complications
Postoperative mortality | Upto one month after hospital discharge
  Death due to surgical complication

CONTACTS AND LOCATIONS:
Overall Officials: Birendra K Sah, PH D, Principal Investigator — Ruijin Hospital; Chen Li, PH D, Study Director — Ruijin Hospital; Zhenggang Zhu, PH D, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanhgai, China

REFERENCES:
- [Derived] Sah BK, Xu W, Zhang B, Zhang H, Yuan F, Li J, Liu W, Yan C, Li C, Yan M, Zhu Z. Feasibility and Safety of Perioperative Chemotherapy With Fluorouracil Plus Leucovorin, Oxaliplatin, and Docetaxel for Locally Advanced Gastric Cancer Patients in China. Front Oncol. 2021 Jan 18;10:567529. doi: 10.3389/fonc.2020.567529. eCollection 2020. PMID 33537232